CLINICAL TRIAL: NCT04237649
Title: A Phase I/Ib, Open-label, Multi-center, Study of KAZ954 as a Single Agent and in Combination With Spartalizumab, NZV930 and NIR178 in Patients With Advanced Solid Tumors
Brief Title: KAZ954 Alone and With PDR001, NZV930 and NIR178 in Advanced Solid Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CKAZ954A12101; 2019-002841-39 (EudraCT Number)
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; KAZ954; PDR001; Spartalizumab; NIR178; NZV930; Immunotherapy; Phase I/Ib
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): KAZ954
  Interventions: Drug: KAZ954
- Arm B (Experimental): KAZ954 + PDR001
  Interventions: Drug: KAZ954; Drug: PDR001
- Arm C (Experimental): KAZ954 + NIR178
  Interventions: Drug: KAZ954; Drug: NIR178
- Arm D (Experimental): KAZ954 + NZV930
  Interventions: Drug: KAZ954; Drug: NZV930

INTERVENTIONS:
Drug: KAZ954 — KAZ954 will be administered in every arm.
Drug: PDR001 — KAZ954 + PDR001
  Arms: Arm B
Drug: NIR178 — KAZ954 + NIR178
  Arms: Arm C
Drug: NZV930 — KAZ954 + NZV930
  Arms: Arm D

SUMMARY:
The primary objective of the trial was to characterize the safety, tolerability, and maximum tolerated dose (MTD)/recommended dose (RD) for expansion of single agent KAZ954 and KAZ954 in combination with PDR001, NIR178 and NZV930.

DETAILED DESCRIPTION:
The purpose of this trial was to explore the clinical utility of several therapies in patients with advanced cancer.

This is a multi-center, open-label Phase I/Ib study. The study consisted of a dose escalation part and a dose expansion part testing KAZ954 as a single agent or KAZ954 in combination with PDR001, NZV930 and NIR178.

The dose escalation part estimated the MTD and/or RD and tested different dosing schedules. The dose escalation arm KAZ954 + NZV930 was not opened.

The dose expansion part of the study was planned to use the MTD/RDE determined in the dose escalation part to assess the activity, safety and tolerability of the investigational products in patients with specific types of cancer. The dose expansion part of the study was not started.

ELIGIBILITY:
Inclusion Criteria:

Patients with metastatic and/or advanced malignancies not amenable to curative treatment by surgery.

Must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening and during the study.

ECOG Performance Status of <2.

Exclusion Criteria:

Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require concurrent treatment - including surgery, radiation and/or corticosteroids.

History of severe hypersensitivity reaction to any ingredient of study drug(s) and other mAbs and/or their excipients.

Impaired cardiac function HIV Known history of tuberculosis Systemic chronic steroid therapy

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 35 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the DLT period. The DLT period for Schedule 1 is 28 days and covers two infusions. The DLT period for Schedule 2 and Schedule 3 is 35 days to cover two infusions of the Experimental dose. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Incidence of adverse events and serious adverse events during the on-treatment period | Up to approximately 52 weeks (KAZ954 single agent), 20 weeks (KAZ954+PDR001) and 24 weeks (KAZ954+NIR178)
  Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs. The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Number of participants with dose interruptions and dose reductions | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  Number of participants with at least one dose interruption or reduction of KAZ954 and its combination partners during study treatment to assess tolerability.
Dose intensity of study treatment | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  Dose intensity of KAZ954 and its combination partners computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per RECIST v1.1 | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  ORR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1. For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Overall Response Rate (ORR) per iRECIST | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  ORR is the percentage of patients with a best overall response of complete response (iCR) or partial response (iPR), based on local investigator assessment per immune-related RECIST (iRECIST). For iRECIST, the principles used to determine objective tumor response are largely unchanged from RECIST v1.1, while the major change of iRECIST is the concept of 'resetting the bar' if RECIST v1.1 progression is followed by tumor shrinkage. Unlike RECIST v1.1, iRECIST requires the confirmation of progression.
Disease Control Rate (DCR) per RECIST v1.1 | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  DCR is the percentage of patients with a best overall response of complete response (CR), partial response (PR) or stable disease (SD), based on local investigator assessment per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1. For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression.
Disease Control Rate (DCR) per iRECIST | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  DCR is the percentage of patients with a best overall response of complete response (iCR), partial response (iPR), stable disease (iSD), based on local investigator assessment per immune-related RECIST (iRECIST). For iRECIST, the principles used to determine objective tumor response are largely unchanged from RECIST v1.1, while the major change of iRECIST is the concept of 'resetting the bar' if RECIST v1.1 progression is followed by tumor shrinkage. Unlike RECIST v1.1, iRECIST requires the confirmation of progression.
Progression-Free Survival (PFS) per RECIST v1.1 | Up to approximately 52 weeks (KAZ954 single agent), 20 weeks (KAZ954+PDR001) and 24 weeks (KAZ954+NIR178)
  For assessment per RECIST v1.1, PFS is the time from date of start of treatment to the date of event defined as the first progression or death due to any cause. If a subject had not had an event, PFS was censored at the date of last adequate tumor assessment. PFS was analyzed using the Kaplan-Meier method.
Progression-Free Survival (iPFS) per iRECIST | Up to approximately 52 weeks (KAZ954 single agent), 20 weeks (KAZ954+PDR001) and 24 weeks (KAZ954+NIR178)
  For assessment per iRECIST, iPFS is the time from date of start of treatment to the date of event defined as the first documented confirmed progression or death due to any cause. If a subject had not had an event, iPFS was censored at the date of last adequate tumor assessment. PFS was analyzed using the Kaplan-Meier method.
Maximum observed serum concentration (Cmax) of KAZ954 | Cycle 1 Day 1 (C1D1) and Cycle 3 Day 1 (C3D1): pre-dose, 1, 24, 72, 168, 240 and 360 hours after the end of the infusion. The duration of the infusion was 2 hours. One cycle=28 days
  Pharmacokinetic (PK) parameters were calculated based on free KAZ954 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Maximum observed serum concentration (Cmax) of PDR001 | Cycle 1 Day 1 (C1D1) and Cycle 3 Day 1 (C3D1): pre-dose, 1, 168, 336 and 672 hours after the end of the infusion. The duration of the infusion was 30 minutes. One cycle=28 days
  PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Maximum observed plasma concentration (Cmax) of NIR178 and its metabolite NJI765 | Cycle 1 Day 1 (C1D1) and Cycle 2 Day 1 (C2D1): pre-dose, 15 minutes, 1, 2, 4 and 6 hours after morning dose and 12 hours after evening dose. One cycle=28 days
  PK parameters were calculated based on NIR178 and NJI765 plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Area under the serum concentration-time curve from time zero to 14 days post dose (AUC0-14d) of KAZ954 | Cycle 1 Day 1 (C1D1) and Cycle 3 Day 1 (C3D1): pre-dose, 1, 24, 72, 168, 240 and 360 hours after the end of the infusion. The duration of the infusion was 2 hours. One cycle=28 days
  PK parameters were calculated based on free KAZ954 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for area under the curve (AUC) calculation.
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) of PDR001 | Cycle 1 Day 1 (C1D1) and Cycle 3 Day 1 (C3D1): pre-dose, 1, 168, 336 and 672 hours after the end of the infusion. The duration of the infusion was 30 minutes. One cycle=28 days
  PK parameters were calculated based on PDR001 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation.
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) of NIR178 and its metabolite NJI765 | Cycle 1 Day 1 (C1D1) and Cycle 2 Day 1 (C2D1): pre-dose, 15 minutes, 1, 2, 4 and 6 hours after morning dose and 12 hours after evening dose. One cycle=28 days
  PK parameters were calculated based on NIR178 and NJI765 plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation.
Number of participants with anti-KAZ954 antibodies | Baseline (before first dose) and post-baseline (assessed throughout the treatment, up to approximately 48 weeks, 16 weeks and 20 weeks for KAZ954 single agent, KAZ954+PDR001 and KAZ954+NIR178, respectively)
  KAZ954 immunogenicity was evaluated in serum samples. Patient anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: ADA-negative sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-reduced ADA-positive: ADA-positive sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-induced ADA-positive: ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive: ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
Number of participants with anti-PDR001 antibodies | Baseline (before first dose) and post-baseline (assessed throughout the treatment, up to approximately 16 weeks)
  PDR001 immunogenicity was evaluated in serum samples. Patient anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: ADA-negative sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-reduced ADA-positive: ADA-positive sample at baseline and at least 1 post-baseline sample, all of which are ADA-negative samples
  * Treatment-induced ADA-positive: ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive: ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
Overall Response Rate (ORR) using RECIST v1.1 and iRECIST by PD-L1 expression | Up to approximately 48 weeks (KAZ954 single agent), 16 weeks (KAZ954+PDR001) and 20 weeks (KAZ954+NIR178)
  Programmed Death-Ligand 1 (PD-L1) expression was assessed centrally using the 22C3 PharmDx assay. PD-L1 expression levels were defined based on the tumor proportion score (TPS). The PD-L1 expression levels were categorized as high (TPS ≥ 50%), medium (TPS 1% - 49%) and low (TPS <1%) expressors. ORR using RECIST v1.1 and iRECIST was summarized by PD-L1 expression.
Progression Free Survival (PFS) using RECIST v1.1 and iRECIST by PD-L1 expression | Up to approximately 52 weeks (KAZ954 single agent), 20 weeks (KAZ954+PDR001) and 24 weeks (KAZ954+NIR178)
  Programmed Death-Ligand 1 (PD-L1) expression was assessed centrally using the 22C3 PharmDx assay. PD-L1 expression levels were defined based on the tumor proportion score (TPS). The PD-L1 expression levels were categorized as high (TPS ≥ 50%), medium (TPS 1% - 49%) and low (TPS <1%) expressors. PFS using RECIST v1.1 and iRECIST was summarized by PD-L1 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (5):
  - University Of California LA, Los Angeles, California
  - Yale University Yale Cancer Center, New Haven, Connecticut
  - Northwestern University Med School, Chicago, Illinois
  - WA Uni School Of Med Dept. of Siteman Cancer Center, St Louis, Missouri
  - Uni of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Shatin New Territories, Hong Kong, Hong Kong
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Sunto Gun, Shizuoka, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18199
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2305